CLINICAL TRIAL: NCT01961011
Title: Simultaneous Bilateral Versus Unilateral Carpal Tunnel Release: A Prospective Comparison of Early Pain and Limitations in Activities of Daily Living
Brief Title: Bilateral vs Unilateral CTR
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Daniel Osei, Assistant Professor of Orthopedic Surgery, Washington University School of Medicine
Other Study IDs: 201206073
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: nerve compression, carpal tunnel, clinical decision making
MeSH Terms: conditions — Carpal Tunnel Syndrome; Neuroma; Median Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort #1: Bilateral carpal tunnel release: Cohort #1: Patients undergoing simultaneous bilateral carpal tunnel release for treatment of bilateral carpal tunnel syndrome. Inclusion criteria includes any adult patient indicated for bilateral carpal tunnel release. Exclusion criteria include age less than 18, pregnancy, any protected patient population, and the lack of assistance at home during the early postoperative period.
- Cohort #2: Unilateral carpal tunnel release: Cohort #2: Patients undergoing unilateral carpal tunnel release fir bilateral carpal tunnel syndrome. Patients will chose which hand they wish to have operated on. Patient will plan on undergoing carpal tunnel release on the unoperated side at a later date. Inclusion criteria include any adult patient indicated for unilateral carpal tunnel release. Exclusion criteria include age less than 18, pregnancy, and any protected patient population.

SUMMARY:
Carpal tunnel release is a well accepted treatment for median nerve compression at the wrist. With a prevalence of 50 per 1000, it is the most common compressive neuropathy. With a number of anatomic as well as systemic factors playing a role in the development of carpal tunnel syndrome, it is not surprising that there is a high incidence of bilaterality with this disease. Padua et al. reported that 87% of 266 consecutive cases had signs and symptoms of carpal tunnel syndrome in their contralateral hand.

In patients who have bilateral carpal tunnel syndrome that has not responded to conservative treatment, surgical release is indicated. In such cases, a decision must be made whether to offer bilateral simultaneous surgical release or to stage the two affected hands to allow time to recover from each.

The purpose of this study is to determine the differences in short term disability between having bilateral vs unilateral carpal tunnel release. With better understanding of the way in which patients are impaired, better recommendations may be made on which patients to indicate for simultaneous bilateral procedures and who would benefit from staging procedures, allowing the patient to recover from one hand prior to proceeding to surgery on the other hand.

DETAILED DESCRIPTION:
Carpal tunnel syndrome is the most common compressive neuropathy, occurring in 0.1 to 3% of the population. The incidence is reported to be higher in certain at risk populations. 87% of individuals exhibit bilateral symptoms. In patients who fail conservative treatment, surgery is indicated. To date, it is not know whether patients benefit from undergoing simultaneous or consecutive carpal tunnel release. Some patients express concern that having both hands operated on may make it impossible to perform necessary activities of daily living in the early postoperative period. Other patients express concern that having two surgeries increases their out of pocket cost, their total disability time, and lengthens the amount of time to resolution of preoperative symptoms. One previous study has attempted to characterize the differences in the effect on activities of daily living of these two treatment paradigms. This study was limited by the fact that there was no comparison group to the study cohort.

Cohort #1: Patients undergoing simultaneous bilateral carpal tunnel release. Inclusion criteria includes any adult patient indicated for bilateral carpal tunnel release. Exclusion criteria include age less than 18, pregnancy, any protected patient population, and the lack of assistance at home during the early postoperative period.

Cohort #2: Patients undergoing unilateral carpal tunnel release. Inclusion criteria include any adult patient indicated for unilateral carpal tunnel release. Exclusion criteria include age less than 18, pregnancy, and any protected patient population.

Once a patient has been identified in the clinic the consent process will begin. Consent will be administered by a member of the research team. Being part of this investigation will not change the standard treatment of carpal tunnel syndrome in any way. After surgery, patients will go home and be asked to fill out the Quick DASH, Levine-Katz Severity Score, WHO HPQ, and SF-6D on pre-operatively and at their first post-operative visit. They will also fill out an activities of daily living log that asks the patient to rate on a scale from 1 to 5 how much difficulty he or she has with each task on the list. The patient will return their ADL log to their physician on their first postoperative visit. A final postoperative visit will occur at 1 month. The investigational questionnaires will be filled out one last time at that visit. No long term follow up is required. Patients will be contacted on their first post-operative day to ensure receipt of the daily log, the day prior to the first post operative visit as a reminder to bring the log into clinic, and on the day before their last post-operative visit thanking them for participation in the study. During their final phone call patients will be asked what factors contributed to their decision to proceed or not proceed with undergoing bilateral carpal tunnel release.

ELIGIBILITY:
Inclusion Criteria

- any adult patient indicated for bilateral carpal tunnel release after having failed nonoperative treatment.

Exclusion Criteria

* age less than 18
* pregnancy
* any protected patient population

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to a tertiary care orthopedic practice with bilateral carpal tunnel syndrome
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change in QuickDASH score | 10 days, 30 days
  The QuickDASH is a shortened version of the DASH Outcome Measure. Instead of 30 items, the QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb.

SECONDARY OUTCOMES:
World Health Organization Health and Performance Questionnaire | 30 days
  The WHO HPQ is a self-reported instrument designed to estimate the workplace costs of health problems in terms of reduced job performance, sickness absence, and work-related accidents-injuries.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States